CLINICAL TRIAL: NCT04840719
Title: A Prospective ,Multicenter, Registry Study of RECO in the Endovascular Treatment of Acute Ischemic Stroke
Brief Title: RECO in the Endovascular Treatment of Acute Ischemic Stroke
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Zhongrong Miao, Director, Department of interventional neurology, Beijing Tiantan Hospital
Other Study IDs: KY 2019-080-03
Record Dates: First submitted 2020-11-06; First posted 2021-04-12 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Intracranial Artery Occlusion With Infarction (Disorder)
Keywords: Acute ischemic stroke; endovascular treatment; registry
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: RECO

SUMMARY:
Investigate Reco ® ,the first clot retriever in china as the primary therapyand remedies in the real world.

DETAILED DESCRIPTION:
Endovascular thrombectomy (EVT) is effective and safe for acute ischemic stroke (AIS) caused by large vessel occlusion (LVO) in major clinical trials. Whether the benefit of EVT in randomized trials could be generalized to clinical practice, especially in developing countries, remains unknown. The Registry was established to evaluate the utilization, and subsequent outcomes of EVT treated AIS patients. This study is a multi-center, prospective registry study initiated by researchers, to investigate Reco ® ,the first clot retriever in china as the primary therapyand remedies in the real world.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Diagnosis of acute ischemic stroke
3. Imaging confirmed intracranial large artery occlusion (LVO): intracranial internal carotid artery (ICA T/L), middle cerebral artery (MCA M1/M2), anterior cerebral artery (ACA A1/A2), basilar artery (BA), vertebral artery (VA V4), and posterior cerebral artery (PCA P1);ASPECT or PC-ASPECT ≥ 6
4. Initiation of any type of endovascular treatment (EVT), including intra-arterial thrombolysis, mechanical thrombectomy, angioplasty, and stenting
5. The patient or the patient's legal representative is able and willing to sign the informed consent

Exclusion Criteria:

1. Isolated cervical ICA or VA occlusion;
2. No evidence of LVO on DSA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute ischemic stroke caused by large vessel occlusion and using RECO to receive endovascular treatment.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-05-22 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
Functional independence at 90 days (modified Rankin Scale of 0-2) | [90±7 days after procedure]
  The range of modified Rankin Scale was from 0 to 6. 0-No symptoms;1-No significant disability;2-Slight disability;3-Moderate disability;4-Moderately severe disability;5-Severe disability;6 -Dead.A higher score indicates worse a outcome.
Symptomatic intracranial hemorrhage (sICH) within 12-36 hours after the procedure | 12-36 hours after the procedure
  Heidelberg Bleeding Classification): new intracranial hemorrhage detected by brain imaging associated with ≥4 points total National Institutes of Health Stroke Scale (NIHSS), ≥2 points in one NIHSS category, leading to intubation/ hemicraniectomy/ EVD placement or other major medical/surgical intervention, or absence of alternative explanation for deterioration
Time from symptom onset to recanalization | From the time of symptom onset until the time of of the recanalization of the occluded artery, assessed up to 48 hours
  Minutes

SECONDARY OUTCOMES:
Recanalization rate at the end of the procedure | Immediately after the procedure
  modified thrombolysis in cerebral infarction (mTICI) 2b-3
Recanalization rate after the first attempt | Immediately after the first attempt of endovascular treatment
  mTICI score 2b-3
Changes in NIHSS score immediately after the procedure | within 2 hours after the procedure
  difference between NIHSS score immediately after the procedure and baseline
Changes in NIHSS score 24 hours after the procedure | 24 hours after the procedure
  difference between NIHSS score 24 hours after the procedure and baseline
Changes in NIHSS score 7 days after the procedure or at discharge | 7 days after the procedure or discharge
  difference between NIHSS score 7 days after the procedure or discharge and baseline
EQ-5D 90 days after the procedure | 90±7 days after the procedure
  EQ-5D is a standardized instrument for measuring generic health status. Rated level can be coded as a number 1, 2, or 3, which indicates having no problems for 1, having some problems for 2, and having extreme problems for 3. As a result, a person's health status can be defined by a 5-digit number, ranging from 11111 (having no problems in all dimensions) to 33333 (having extreme problems in all dimensions).A higher score indicates a better outcome.
Barthel index (BI) 90 days after the procedure | 90±7 days after the procedure
  The BI has a score of 0-100. A higher score indicates a better outcome.
Parenchymal hematoma (PH2) | 12-36 hours after the procedure
  PH2 is defined as the rate of hematoma >30percent in infarct area
Any intracranial hemorrhage on imaging | 12-36 hours after the procedure
  Based on the image
All-cause mortality within 90 days | 90±7 days after the procedure
  mortality
Time from onset to arrival | At baseline, after arrival at the hospital immediately
  record the time
Time from arrival to imaging | At baseline, after taking any brain imaging immediately
  record the time
Time from imaging to puncture | At baseline, during the procedure, after successful groin puncture immediately
  record the time
Time from puncture to recanalization | At baseline, during the procedure, after successful recanalization immediately
  record the time

CONTACTS AND LOCATIONS:
Overall Officials: Zhongrong Miao, PhD,MD, Principal Investigator — Capital Medical University, Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ding Y, Zhai T, Chen R, Chen F, Cheng Y, Zhu S, Liu Y, Xiao G, Zhang Y, Liu Y, Miao Z, Niu J. A prospective, multicentre, registry study of RECO in the endovascular treatment of acute ischaemic stroke. Sci Rep. 2024 Jan 25;14(1):2196. doi: 10.1038/s41598-024-52207-z. PMID 38272958